CLINICAL TRIAL: NCT07310901
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Dose-Range Finding Study of the Efficacy, Safety, and Pharmacokinetics of CRB-913 in Participants With Obesity With a Single Cohort Open-label Exploratory Pharmacokinetic Lead-In
Brief Title: A 2-part, Phase 1b Clinical Study Designed to Evaluate the Safety, PK, and Efficacy of CRB-913 in Participants With Obesity
Acronym: CANYON-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRB-913-02
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Obese But Otherwise Healthy Participants
Keywords: Obesity; Body Weight; Nutritional and Metabolic Diseases; Metabolic Diseases; Endocrine System Diseases; Overweight; Nutrition Disorders; Cannabinoid-1 receptor inverse agonist
MeSH Terms: conditions — Obesity; Body Weight; Nutritional and Metabolic Diseases; Metabolic Diseases; Endocrine System Diseases; Overweight; Nutrition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 is open label. Part 2 is double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: PK Lead-in (Experimental): Primary Treatment Period (Day 1): Participants will receive a single dose of CRB-913. Following Part 1 of the study Part 2 will open for recruitment.
  Safety Follow-up Period: Participants who complete or discontinue the primary treatment period are followed for safety for 28 days. No treatment is administered during this period.
  Interventions: Drug: CRB-913
- Part 2: CRB-913 low dose (Experimental): Primary Treatment Period (Day 0-Day 85): Participants will receive CRB-913 low dose which is maintained up to day 85.
  Safety Follow-up Period: Participants who complete or discontinue the primary treatment period are followed for safety for 28 days. No treatment is administered during this period.
  Interventions: Drug: CRB-913
- Part 2: CRB-913 Medium Dose (Experimental): Primary Treatment Period (Day 0-Day 85): Participants will receive CRB-913 starting at low dose for 14 days and increasing to medium dose at day 15 which is maintained up to day 85.
  Safety Follow-up Period: Participants who complete or discontinue the primary treatment period are followed for safety for 28 days. No treatment is administered during this period.
  Interventions: Drug: CRB-913
- Part 2: CRB-913 High Dose (Experimental): Primary Treatment Period (Day 0 - Day 85): Participants will receive CRB-913 starting at low dose for 14 days, increasing to medium dose at day 15 for 14 days and then increased to high dose at day 29 which is maintained up to day 85.
  Safety Follow-up Period: Participants who complete or discontinue the primary treatment period are followed for safety for 28 days. No treatment is administered during this period.
  Interventions: Drug: CRB-913
- Part 2: Placebo (Placebo Comparator): Primary Treatment Period (Day 0-Day 85): Participants will receive CRB-913 matching placebo which is maintained up to day 85.
  Safety Follow-up Period: Participants who complete or discontinue the primary treatment period are followed for safety for 28 days. No treatment is administered during this period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRB-913 — Administered QD
  Arms: Part 1: PK Lead-in; Part 2: CRB-913 High Dose; Part 2: CRB-913 Medium Dose; Part 2: CRB-913 low dose
Drug: Placebo — Administered QD
  Arms: Part 2: Placebo

SUMMARY:
This study will assess the safety of the investigational drug CRB-913 and how it is processed in the body.

The study has two parts: Part 1 will measure drug levels in healthy adults after taking CRB-913 tablets, and Part 2 will compare three doses of CRB-913 with placebo to evaluate safety, effects on body weight, and drug levels in the blood.

Part 2 is blinded, meaning participants, study doctors, and the sponsor will not know which treatment is given.

Participants in Part 2 will take study treatment for 12 weeks and will be followed for 28 days after treatment ends.

DETAILED DESCRIPTION:
CRB-913 is a novel cannabinoid receptor type 1 (CB1) inverse agonist (CB1-IA) that is being developed for once-daily treatment of obesity.

This study will look at how the investigational drug CRB-913 behaves in the body and how it affects body weight.

The study has two parts:

Part 1 will include healthy adult participants. They will receive CRB-913 in tablet form. Researchers will measure how much of the drug enters the bloodstream and how long it stays there.

Part 2 will include participants who will receive one of three different doses of CRB-913 or a placebo (a tablet with no active drug). This part of the study will look at the safety of CRB-913 and its effects on body weight. Researchers will also measure the amount of CRB-913 in the blood.

Part 2 is blinded, which means that participants, study doctors, and the study sponsor will not know who is receiving CRB-913 or placebo.

All participants in Part 2 will take their assigned study tablets for 12 weeks, followed by a 28-day follow-up period after treatment ends.

The information collected in this study will help determine whether CRB-913 is safe, how the body processes it, and whether it may help with weight-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Participants with BMI 18.0-25.0 kg/m²
* Part 2: Obese participants with BMI ≥30 kg/m²

Exclusion Criteria:

* Significant liver disease or moderate-severe hepatic impairment
* History of seizures, epilepsy, or intracranial surgery
* Diabetes mellitus (Type 1 or Type 2), except gestational
* Bariatric surgery or >5 kg weight change in past 3 months
* Recent use (within 3 months) of GLP-1 agonists or other weight-loss medications
* Major depression within 2 years.
* Any history of suicidal ideation/attempt
* Severe psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* Elevated screening scores: PHQ-9 >4, GAD-7 >4, or positive C-SSRS Items 1-2
* Active or recent (within 5 years) malignancy (exceptions: in situ and fully resected nonmelanoma skin cancer)
* Abnormal thyroid function: TSH >6 mIU/L unless stable on replacement therapy
* QTc >470 msec (females) or >450 msec (males) or history of long QT syndrome
* Use of systemic corticosteroids or unstable chronic medications affecting BP, lipids, or glucose
* Use of CYP3A4 substrates or strong P-gp substrates/inhibitors
* Investigational drug use within 28 days
* Prior exposure to CRB-913 or other CB1 inverse agonists/antagonists
* Substance abuse history
* Pregnancy, breastfeeding, or unwillingness to use highly effective contraception
* Positive drug or alcohol screen
* Any condition that, in the investigator's judgment, makes participation unsafe or non-feasible

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: To evaluate the PK of a single dose of CRB-913 - Cmax | 0 to 48 hours
  Maximum plasma concentration (Cmax)
Part 1: To evaluate the PK of a single dose of CRB-913 - Tmax | 0 to 48 hours
  Time to maximum plasma concentration (Tmax)
Part 1: To evaluate the PK of a single dose of CRB-913 - T1/2 | 0 to 48 hours
  Terminal elimination half-life (T1/2)
Part 2: To evaluate the safety of CRB-913 - TEAE | Day 1 to 28 days post final dose
  Incidence and severity of treatment emergent adverse events
Part 2: To evaluate the safety of CRB-913 - AESI | Day 1 to 28 days post final dose
  Incidence of adverse events of special interest

SECONDARY OUTCOMES:
Part 1: To evaluate the safety of a single dose of CRB-913 - TEAE | Day 1 to 28 days post final dose
  Incidence and severity of treatment emergent adverse events
Part 2: To evaluate the effect of CRB-913 on weight | Day 1 to 28 days post final dose
  Mean change in absolute body weight from baseline to End of Treatment (EOT) compared to placebo
Part 2: To evaluate the PK of CRB-913 - Cmax | Day 1 to 28 days post final dose
  Maximum plasma concentration (Cmax)
Part 2: To evaluate the PK of CRB-913 - Tmax | Day 1 to 28 days post final dose
  Time to maximum plasma concentration (Tmax)

OTHER OUTCOMES:
Part 2: To evaluate changes in food noise | Day 1 to 28 days post final dose
  Mean change from baseline in food noise questionnaire (FNQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace Clinical Pharmacology
Locations (15):
- United States (15):
  - Central Alabama Research, Birmingham, Alabama
  - Arizona Clinical Trials, Chandler, Arizona
  - Prospective Research Innovations, Rancho Cucamonga, California
  - Accel Research Sites, DeLand, Florida
  - Tampa Bay Medical Research, Largo, Florida
  - Quotient Sciences, Miami, Florida
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Alliance Clinical, Las Vegas, Nevada
  - Neurobehavioral Research, Cedarhurst, New York
  - Rochester Clinical Research, Rochester, New York
  - Lucas Research, Morehead City, North Carolina
  - Medpace Clinical Pharmacology, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Ohio
  - Velocity Clinical Research, Dallas, Texas
  - Flourish Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided